CLINICAL TRIAL: NCT04513821
Title: CITI-100 EA - Intermediate-Size Expanded Access, Open-Label Study for Use of Mino-Lok Therapy (MLT) in Combination With Systemic Antibiotics in the Treatment of Central Line Associated Bloodstream Infection
Brief Title: Expanded Access: Mino-Lok Therapy (MLT) for the Treatment of CRBSI/CLABSI
Acronym: MLK
Status: Available | Type: Expanded Access
Sponsor: Leonard-Meron Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CITI-100 EA
Record Dates: First submitted 2020-08-10; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections | interventions — Standard of Care; Edetic Acid; Ethanol

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Mino-Lok Therapy (MLT) — Standard of Care antibiotics appropriate for the infecting organism plus Mino-Lok therapy to disinfect and save the catheter. Mino-Lok is made available through this expanded access protocol to patients who otherwise do not qualify for the phase 3 clinical trial (NCT02901717) Other Name: Standard of care antibiotics + Mino-Lok
  Other Names: Standard of care plus MLT. MLT contains minocycline with EDTA and ethanol.

SUMMARY:
This is an Intermediate-Size Expanded Access, Open-Label Study for Use of Mino-Lok Therapy (MLT) in Combination with Systemic Antibiotics in the Treatment of Central Line Associated Bloodstream Infection. Mino-Lok may be made available for patients who otherwise do not qualify for the phase 3 clinical trial (NCT02901717 )

DETAILED DESCRIPTION:
This is an Intermediate-Size Expanded Access, Open-Label Study for Use of Mino-Lok Therapy (MLT) in Combination with Systemic Antibiotics in the Treatment of Central Line Associated Bloodstream Infection.

Mino-Lok Therapy is being developed as an adjunctive therapy for the treatment of catheter-related or central line associated bloodstream infection (CRBSI/CLABSI) in combination with appropriate systemic antibiotic(s), to preserve central venous access and to avoid the complications and morbidities associated with catheter removal and reinsertion.

This is an expanded access program (EAP). This program is designed to provide access to Mino-Lok. A physician must decide whether the potential benefit outweighs the risk of receiving an investigational therapy.

To learn more about this study, please refer to this study by its ClinicalTrials.gov identifier (NCT number): NCT02901717

ELIGIBILITY:
Inclusion Criteria:

1. Subject or a legally authorized representative must provide a signed informed consent form;
2. The subject should be male or female at least 12 years of age. This product has not been studied in a younger pediatric population;
3. Subject should have a bloodstream infection with no other apparent source other than the CVC that meets one of the following criteria:

   * A recognized single pathogen cultured from 1 or more blood cultures; OR
   * A common skin contaminant cultured from 2 or more blood cultures drawn on the same or consecutive calendar days from a subject with fever (>38.0 C), chills, or hypotension (systolic blood pressure <90 mmHg); Note that these criteria are based on the CDCs definition of CLABSI. Please consult the CDC website for guidance at https://www.cdc.gov/nhsn/pdfs/pscmanual/4psc_clabscurrent.pdf.
4. Subjects for whom, in the Investigator's opinion, catheter retention is reasonable or required;
5. This product has not been studied in women who are pregnant or lactating. It's effect on sperm development has also not been studied. Please consider this with female patients that are pregnant or who plan to become pregnant, or female patients who are breastfeeding. Likewise, male patients should refrain from sperm donation for 90 days following exposure to MLT. NOTE: Highly effective methods of contraception include hormonal contraceptives, intrauterine device, double-barrier method, partner sterility, or abstinence are strongly recommended.

Exclusion Criteria:

Subjects who meet any of the following criteria should not be exposed to MLT:

1. Subjects with hypersensitivity or allergy to tetracycline antibiotics or edetate disodium;
2. Subjects taking disulfiram at the time of enrollment or who are expected to take disulfiram at any time during treatment with study drug;
3. The benefit of MLT in subjects with prosthetic cardiac valves, vascular grafts, pacers, automatic implantable cardioverter-defibrillator, or other non-removable vascular foreign body should be evaluated prior to exposure. The Investigator should be confident that these are not the source of infection;
4. The benefit of MLT in subjects with a deep-seated intravascular source of infection (eg, endocarditis [as evidenced by vegetations on an echocardiogram or clinical suspicion] or septic thrombosis) should be evaluated prior to exposure. The Investigator should be confident that these are not the source of infection.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (30):
- United States (27):
  - Phoenix VA Health Care System, Phoenix, Arizona
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida - Shands Hospital - Dialysis Center, Gainesville, Florida
  - Edward Hines Jr. VA Hospital, Hines, Illinois
  - AMG Oncology, Park Ridge, Illinois
  - Lutheran Hospital, Park Ridge, Illinois
  - Indiana Blood and Marrow Institute, Indianapolis, Indiana
  - Ascension Via Christi Hospital, Wichita, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Vincent Hospital, Worcester, Massachusetts
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Health Systems, Detroit, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - VA Sierra Nevada Health Care Systems, Reno, Nevada
  - Saint Michael's Medical Center, Newark, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Carolinas Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Salem VA Medical Center, Salem, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Puerto Rico (3):
  - VA Caribbean Healthcare System, San Juan, PR
  - Manati Medical Center, Manatí
  - Ponce Research Institute, Ponce